CLINICAL TRIAL: NCT01262170
Title: A Randomized, Double-Blind, Active-Controlled, Crossover, Pilot Study to Evaluate the Safety and Efficacy of CigRx™ Lozenge, a Non-Nicotine Non-Tobacco Dietary Supplement, in Daily Smokers in Temporarily Reducing the Desire to Smoke
Brief Title: A Pilot Study to Evaluate Safety and Efficacy of CigRx™ in Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rock Creek Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCP-002
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Smoking; Tobacco Use Disorder
Keywords: dietary supplement; nutraceutical
MeSH Terms: conditions — Smoking; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CigRx Lozenge (Experimental): CigRx Lozenge
  Interventions: Dietary Supplement: CigRx Lozenge
- Tobacco Lozenge (Active Comparator): Tobacco Lozenge
  Interventions: Other: Tobacco Lozenge

INTERVENTIONS:
Dietary Supplement: CigRx Lozenge — lozenge made of dietary supplements
  Arms: CigRx Lozenge
Other: Tobacco Lozenge — lozenge made of compressed cured tobacco extract
  Arms: Tobacco Lozenge

SUMMARY:
A randomized, double-blind, active-controlled, crossover, pilot study to evaluate the safety and efficacy of CigRx™ Lozenge, a dietary supplement, in daily smokers in temporarily reducing the desire to smoke

DETAILED DESCRIPTION:
Subjects will orally self-administer 2 study products, each in the form of a dissolvable lozenge, and will complete questionnaires on demographics, urges to smoke, and product rating.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult smokers
* Smoking for at least 5 years
* Smoking at least one (1) pack of cigarettes a day

Exclusion Criteria:

* Allergy to lozenge components

Ages: 23 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Effect on subject's craving to smoke | 4 hours
  craving is assessed by changes in questionnaire answers over time

SECONDARY OUTCOMES:
Collection of information on adverse events related to study products | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Maria Varga, MD, Principal Investigator — Star Scientific, Inc
Locations (1):
- Comfort Inn, Martinsburg, West Virginia, United States